CLINICAL TRIAL: NCT07294768
Title: Mechanical Power-Guided Lung Protective Ventilation (VentCoach) in Acute Hypoxemic and/or Hypercapnic Respiratory Failure: A Feasibility, Double Arm, Single-blinded Study
Brief Title: Mechanical Power-Guided Lung Protective Ventilation (VentCoach) in Acute Hypoxemic and/or Hypercapnic Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gustavo A. Cortes Puentes, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-004855
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Mechanical Ventilation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Patients randomized to the standard of care group will continue to receive ventilator management per the ARDSnet-based protocol
  Interventions: Other: Standard of Care
- VentCoach (Experimental): Patients randomized to the VentCoach group, in addition to the standard of care, will also receive intermittent ventilator setting adjustments per the VentCoach protocol
  Interventions: Other: VentCoach; Other: Standard of Care

INTERVENTIONS:
Other: VentCoach — VentCoach, a mechanical power-guided lung protective ventilation protocol, will be used to set ventilator adjustments.
  VentCoach ventilator assessments and adjustments will be performed within one hour after enrollment, and then every 4 hours thereafter
  Arms: VentCoach
Other: Standard of Care — Intubated patients will be managed per the standard of care ARDSnet-based mechanical ventilation management at Mayo Clinic, with routine RT/MD assessments, and ventilator setting changes as necessary for the treatment of the patient.

SUMMARY:
The purpose of this research is to evaluate a different way of using the mechanical ventilator device to help better protect the lungs while the patient recovers. We will compare VentCoach to the current standard mechanical ventilation techniques used in our Intensive Care Units.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute hypoxemic and/or hypercapnic respiratory failure.
* Patients requiring intubation and mechanical ventilation for more than 24 hours.
* VentCoach protocol is specific to volume controlled continuous mandatory ventilation (S-CMV).
* Patient who are admitted to RMH 10-3/10-4 and MB 6BGF ICUs.
* Age greater than or equal to 18 years.
* Patient's legal representative should be able to provide informed consent to the study. Any participant speaking any language will be offered participation.

Exclusion Criteria:

* Intubation and mechanical ventilation for airway protection in the setting of procedures/surgeries, e.g. interventional radiology, surgery, or endoscopy.
* Intubation and mechanical ventilation due to drug overdose with expected extubation of less than 24 hours.
* Intubation and mechanical ventilation in the setting of cardiac arrest.
* Intubation and mechanical ventilation for a primary neurological etiology, e.g. increased intracranial pressure, tumor mass effect, ischemic/hemorrhagic stroke, status epilepticus, etc.
* Mechanical ventilation to be guided by esophageal balloon.
* Subject deprived of freedom, minor, subject under a legal protective measure.
* Change in end-of-life decision anticipated after enrollment (or estimated 6-month mortality rate of greater than 50%).

Note: prone positioning is not a contraindication for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Adherence to the VentCoach protocol | 1 year
  Total number of patients to achieve adherence will be defined as documented reduction in mechanical power (MP) or MP less than 12 J/min, in the 16 patients assigned to the VentCoach group

SECONDARY OUTCOMES:
Time to removal from ventilator | 1 year
  Time to successful extubation, allocation to ECMO, or death reported in number of days
Incidence of patient-ventilator dyssynchrony | 1 year
  Number of patients to experience patient-ventilator dyssynchrony, defined as double triggering and flow starvation
Overall use of sedation | 1 year
  Total use of analgesia, converted to morphine equivalent
Overall use of paralytics | 1 year
  Total number of patients to require paralytics: bolus and infusion of neuromuscular blockade outside intubation procedure
Oxygenation index | Baseline, end of treatment (up to 14 days)
  Oxygenation index is calculated by the following equation: mean airway pressure MAP (in cmH2O) × FiO2 × 100 ÷ PaO2 and is reported as a single number.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo A. Cortes Puentes, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20555865